CLINICAL TRIAL: NCT04196582
Title: Comparison of LMA® Gastro Airway and Gastro-Laryngeal Tube in Endoscopic Retrograde Cholangiopancreatography: a Prospective Randomized Observational Trial
Brief Title: LMA® Gastro Airway Versus Gastro-Laryngeal Tube in Endoscopic Retrograde Cholangiopancreatography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Harun UYSAL, Anesthesiology And Reanimation Specialist, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bezmialem Vakif University
Record Dates: First submitted 2019-11-25; First posted 2019-12-12 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Supraglottic Airway Efficiency; Airway Complication of Anesthesia; Airway Aspiration; Complication of Anesthesia; Esophagus Injury; Endoscopic Ergonomics; ERCP Airway Management
Keywords: LMA gastro airway; Gastro-laryngeal tube; ERCP; airway complications

STUDY DESIGN:
Who Masked: Participant
Masking Description: closed envelope.technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastro-laryngeal tube Group (Group G) (Active Comparator): Patients wear Gastro-laryngeal tube after receiving general anesthesia for biliopancreatic procedures
  Interventions: Device: Comparison of LMA Gastro Airway® and Gastro-Laryngeal Tube in patients who will undergo biliopancreatic procedures.
- LMA Gastro Airway Group (Group L) (Active Comparator): Patients wear LMA Gastro Airway® after receiving general anesthesia for biliopancreatic procedures
  Interventions: Device: Comparison of LMA Gastro Airway® and Gastro-Laryngeal Tube in patients who will undergo biliopancreatic procedures.

INTERVENTIONS:
Device: Comparison of LMA Gastro Airway® and Gastro-Laryngeal Tube in patients who will undergo biliopancreatic procedures. — comparing efficiency and complications of second generation airway devices which can use for gastrointestinally procedures

SUMMARY:
Comparison of second generation supraglottic airway devices about anesthesiologist, endoscopist and patient, which used for gastrointestinal procedures. The investigators believe that the endoscope will be easier to reach by the part of GLT extending to the esophagus, but the structural stiffness of this part may damage the esophageal mucosa. On the other hand, since the endoscopic canal of the LMA® Gastro ends at the upper end of the esophagus, it may be more difficult to orient the endoscope to the esophagus, but it may be superior in terms of ventilation efficiency. Therefore these two device worth for comparing.

DETAILED DESCRIPTION:
Supraglottic airway (SGA) devices are produced for avoiding endotracheal intubation for anesthesic interventions. Second generation SGA's like GLT and LMA® Gastro airway are using for endoscopic biliopancreatic procedures. Both of them have an airway canal and endoscopic canal. Although they can use for same reason, their designs are different. So, their airway securities, endoscopic manipulations and complications, would be different.

This study planned as single blind. American Society of Anesthesiologists (ASA) Physical status 1-2 100 patients which will be take endoscopic retrograde cholangiopancreatography (ERCP) included. The study starts after randomization and ends after discharge from the recovery room. All patients will be monitorised for hemodynamic parameters. Depth of anesthesia will be provided by bispectral index (BIS) monitoring. After anesthesia induction SGA will placed by an experienced anesthesiologist. Bilateral chest movements and auscultation, capnogram graphy and oropharyngeal leak pressure test will be used for confirmation of placement. After procedure endoscopist will take pictures of esophagus and hypopharynx. After extubation and sufficient consciousness and breathing of patient, patients will be transferred to post-anaesthesia care unit (PACU). Vital parameters will continue to monitoring in PACU. Patients will be discharge as usual with an Aldrete score ≥ 9.

Data will be collected during the procedure and in recovery room. Data will be stored in electronic database without mention to patient's name.

ELIGIBILITY:
Inclusion Criteria:

* ASA Physical Status 1-2
* Elective Procedures
* Weight 50-100 Kg

Exclusion Criteria:

* Laryngeal mask airway contraindications.
* Anesthesic drug allergies
* Height <155 cm
* Body Mass index > 35 kg/m2
* Alcohol or narcotic drug usage
* Restrictive or obstructive pulmonary diseases
* Hepatic cardiac or renal failure
* Psychotic problems
* Neurologic or cognitive deficiencies.
* Pregnancy
* Difficult airway or facial deformities
* Previous cervical surgery or cervical radiotherapy
* Previous esophagus surgery
* High risk of pulmonary aspiration

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-07-10 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | Intra-operative; after device insertion
  Oropharyngeal leak pressure is the airway pressure at which the circuit pressure stabilizes by closing the expiratory valve of the circle system at a constant gas flow of 3 L / min.
Endoscopist satisfaction analysis: score | Immediately after the procedure
  Endoscopist will score from 0 (worst) to 10 (best)
Leakage rate percentages | Intra-operative; after device insertion at first minute
  The leakage rate percentage is the calculation of the difference between the adjusted tidal volume and the exhaled tidal volume and then proportioning to the adjusted tidal volume.

SECONDARY OUTCOMES:
Hypopharyngeal/Esophageal Mucosal status | Within the first minute after the procedure is completed, while the duodenoscope is being removed while it passes through the esophagus and hypopharynx
  Number of patients with hyperemia, laceration (while extubating patient, endoscopist will take pictures of esophagus for if there is any mucosal damage). Esophageal and hypopharyngeal mucosal damage was determined in 5 grades by a visual mucosal damage scoring system [grade 1- normal mucosa, grade 2- mild hyperemia, grade 3-severe hyperemia, grade 4-bloody gross hyperemia, grade 5- laceration].
Blood staining on the device | Immediately after removing the supraglottic airway device
  Whether there is blood on the supraglottic airway device or not
Presence of sore throat | One hour after extubation
  Sore throat if present, was classified as mild, moderate or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)